CLINICAL TRIAL: NCT00078598
Title: A Multi-Center, Randomized, Phase III Study of Rituximab Versus Iodine I 131 Tositumomab Therapy for Patients With Relapsed Follicular Non-Hodgkin's Lymphoma
Brief Title: A Study of Rituximab Versus Iodine I 131 Tositumomab Therapy for Patients With Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corixa Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCBX001-049
Record Dates: First submitted 2004-03-01; First posted 2004-03-03 (Estimated); Last update posted 2005-11-09 (Estimated); Status verified 2004-10

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Relapsed; Follicular
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — Rituximab

INTERVENTIONS:
Drug: Rituximab or Iodine I 131 Tositumomab Therapy

SUMMARY:
A total of 506 patients, 253 per arm, will be enrolled at 30 to 40 sites in the United States and Europe.

Patients will be randomly assigned to one of two treatment arms. In Arm A, patients will receive 375 mg/m2 of rituximab (US, Canada - Rituxan®; EU - Mabthera®), given as an IV infusion once weekly for 4 weeks. In Arm B, patients will receive Iodine I 131 Tositumomab therapy. For Arm B, patients undergo a two-phase treatment. In the first phase, termed the "dosimetric dose," patients will receive an infusion of unlabeled Tositumomab (450 mg) immediately followed by an infusion of Tositumomab (35 mg) that has been labeled with 5 mCi (0.18 GBq) of iodine 131. Whole body gamma camera scans will be obtained three times (Day 0, Day 2, 3, or 4, and Day 6 or 7) following the dosimetric dose. Using the dosimetric data from these three imaging timepoints, the patient's weight, and platelet count, a patient-specific administered activity of iodine I 131 Tositumomab (expressed in mCi or GBq) will be calculated to deliver the desired total body dose of radiation (65 or 75 cGy). In the second phase, termed the "therapeutic dose," patients in Arm B will receive an infusion of unlabeled Tositumomab (450 mg) immediately followed by an infusion of the patient-specific administered activity of Iodine 131-conjugated Tositumomab (35 mg).

Patients on study will be followed for response and safety at Week 7, Week 13, and every 3 months for the first and second years, every 6 months for the third year, and then annually for the fourth and fifth years. Patients will be followed for safety only annually for years 6-10.

ELIGIBILITY:
Inclusion Criteria

* A histologically confirmed diagnosis of follicular lymphoma, Grade I, II, or III (WHO/REAL Classification) (follicular, small cleaved; follicular, mixed small-cleaved and large-cell; or follicular large-cell lymphoma in the International Working Formulation).
* Recurrent lymphoma after one or two qualifying therapy regimen(s).
* A performance status of at least 70% on the Karnofsky Scale.
* An absolute neutrophil count > 1500 cells/mm3 and a platelet count > 100,000 cells/mm3.
* Adequate renal function and adequate hepatic function.
* Bi-dimensionally measurable disease with at least one lesion measuring > or equal to 2.0 x 2.0 cm (i.e., > 4.0 cm2) by CT scan.
* HAMA negative.
* At least 18 years of age.
* Give written informed consent by signing an IRB/ethics committee approved informed consent form prior to study entry.

Exclusion Criteria

* Histological transformation to diffuse,large cell lymphoma
* More than 1 course of rituximab
* Disease better treated with limited field therapy
* Involvement of >25% of the intratrabecular marrow
* Active infection
* Significant cardiac disease
* Prior ChemoRx, biological therapy, radiation Rx, or high dose systemic steroid therapy within 8 weeks
* Prior radioimmunotherapy
* History of another malignancy
* HBsAg positivity
* CNS involvement with lymphoma
* Pregnant or nursing
* Ascites by physical exam
* Previous use of non-human monoclonal antibody therapy, known hypersensitive to murine proteins
* Hydronephrosis
* Radiotherapy to >25% of the blood forming marrow
* Prior stem cell transplant
* Failed stem cell harvest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506
Dates: Start 2004-04

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Northside Hospital, Atlanta, Georgia
  - Medical Oncology/Hematology Associates, Dayton, Ohio
  - Madigan Army Medical Center, Tacoma, Washington
  - St Mary Medical Center/Regional Cancer Center, Walla Walla, Washington
  - West Virginia University/Mary Babb Randolph Cancer Center, Morgantown, West Virginia